CLINICAL TRIAL: NCT03584126
Title: Imaging-based, Non-invasive Diagnosis of Persistent Atrial Fibrillation - imATFIB
Brief Title: Imaging-based, Non-invasive Diagnosis of Persistent Atrial Fibrillation
Acronym: imATFIB
Status: Completed | Type: Observational
Sponsor: County Clinical Emergency Hospital Cluj-Napoca (Other)
Responsible Party: Sponsor
Other Study IDs: 20117/04.10.2016
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AF: Patients with atrial fibrillation visiting the outpatient clinic; examined by general examination, electrocardiography, ecocardiography and MRI.
  Interventions: Diagnostic Test: Electrocardiography, ecocardiography and MRI.
- Control: Healthy adult volunteers; examined by the study physicians by general examination, electrocardiography, ecocardiography and MRI.
  Interventions: Diagnostic Test: Electrocardiography, ecocardiography and MRI.

INTERVENTIONS:
Diagnostic Test: Electrocardiography, ecocardiography and MRI. — AF patients and healthy adult volunteers will be examined by the study physicians and included in the study according to the inclusion criteria. After a general examination, an electrocardiography, an ecocardiography and an MRI will be performed on the AF-affected and healthy hearts, respectively.

SUMMARY:
The main objective of the present project is to develop an imaging-based tool to determine the origin and cause of persistent atrial fibrillation (AF). The result of the study is a diagnostic method which aids the medical work-up of patients suffering from this disease.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia associated with substantial morbidity and mortality in humans. Histopathological studies of persistent AF have reported extracellular matrix remodeling with fibrotic infiltration which may cause atrial dilation. The degree of the fibrosis might have a significant impact on wave propagation during AF. The main objective of the present project is to develop an imaging-based tool to determine the origin and cause of persistent AF. The obtained clinical parameters of patients and controls (electrocardiography, ecocardiography and MR imaging data) will be correlated with known markers in order to identify novel markers for AF diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-80 years
* weight: 50-120 kg
* persistent, permanent or paroxysmal atrial fibrillation
* clinically stable patients: outside of an acute cardiac event with constant chronic medication
* optimum echographic window

Exclusion Criteria:

* patients with: rheumatic mitral disease; acute myocardial-pericarditis; chronic rheumatism, under chronic or immunomodulatory treatment; infectious-inflammatory process of any cause
* patients undergoing oncology treatment
* patients under medication in another study
* patients undergoing immunosuppressive therapy
* contraindication for magnetic resonance imaging (MRI)
* patients with valvular prosthesis, pacemaker of any type, metallic elements in the body (including metal particles accidentally in the body or as a result of exercising certain professions); pregnant patients; patients with known poly-allergy; patients with altered renal function (creatinine clearance <40 mL/min determined by the Cockcroft-Gault formula).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population presented at the cardiologist with persistent, permanent or paroxysmal atrial fibrillation (AF).
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Correlation of the presence, localization and quantity of left atrial fibrosis assessed by MRI in patients with persistent atrial fibrillation. | 2016-2020
  A. Percentage of patients with left atrial fibrosis assessed by MRI among those with persistent atrial fibrillation.
  B. Correlation of the left atrial fibrosis localization and amount with persistent atrial fibrillation severity.

SECONDARY OUTCOMES:
Specificity of left atrial fibrosis for persistent atrial fibrillation by comparing fibrosis in patients and healthy volunteers. | 2016-2020
  A. Correlation of left atrial fibrosis with left atrial dimensions in patients and healthy volunteers.
  B. Correlation of left atrial fibrosis with blood bio-marker levels and echocardiography parameters in patients and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Bálint, PhD, Principal Investigator — County Clinical Emergency Hospital Cluj-Napoca
Locations (1):
- County Clinical Emergency Hospital of Cluj-Napoca, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manole S, Pintican R, Budurea C, Pop S, Iancu SD, Popa L, Coman M, Schiau C, Coman V, Schiau S, Balint Z. Increased Left Ventricular Mass Index and Atrial Volume Index Are Associated with Atrial Fibrosis in Patients with Atrial Fibrillation. J Clin Med. 2025 Sep 12;14(18):6432. doi: 10.3390/jcm14186432. PMID 41010636